CLINICAL TRIAL: NCT01401400
Title: Genetic Study of Peginterferon Treatment in Hepatitis B Patients: The GIANT-B Study
Acronym: GIANT-B
Status: Completed | Type: Observational
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Other Study IDs: HBV10-03
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood samples from which DNA can be isolated
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- (Peg) interferon: Patients who are treated for at least 12 weeks with (peg-)interferon for chronic hepatitis B

SUMMARY:
Background and rationale Chronic hepatitis B is the most common cause of liver cirrhosis and hepatocellular carcinoma worldwide.(1) Antiviral therapy with oral nucleoside analogs and interferon can reduce viral load and hepatic necroinflammation, and may reduce the risk of hepatocellular carcinoma and cirrhotic complications. (2-4) Peginterferon has both direct antiviral and immunomodulatory effects. The advantages of this drug include a finite course of treatment and the lack of drug resistance. However, it requires subcutaneous injections and carries some side effects. Besides, only 30% to 40% of treated patients have sustained response to treatment.(5-8) To reduce the costs and side effects of treatment, it is important to predict if a patient will respond to peginterferon. Genetic host studies on peginterferon response will provide a lot of knowledge on the interaction between the host and the virus to induce immune control, also outside the setting of immune modifying therapy. Recently, genome wide association studies (GWAS) identified genetic polymorphisms of the IL28B gene that were shown to be associated with treatment response to interferon and ribavirin in patients with chronic hepatitis C.(9-12) The same polymorphisms are also associated with natural clearance of hepatitis C virus. Whether the same phenomenon applies to patients with chronic hepatitis B is unclear. Furthermore, response to conventional interferon has shown to decrease the risk of hepatocellular carcinoma and to prolong survival.(13) Virological and serological response to PEG-IFN is durable in a substantial proportion of patients through 3 years of follow-up (14), but whether treatment benefits are sustained after that period and amount to clinically meaningful results is unknown. To date, a GWAS to predict the response to peginterferon in chronic hepatitis B patients has not been performed. Polymorphisms in genes such as IL28B can be identified through a GWAS and can be used to assess the chance of response to treatment and select patients who have a high probability of response to peginterferon.

We aim to perform a GWAS in chronic hepatitis B patients previously treated with peginterferon to identify polymorphisms in genes that are associated with response to this treatment regimen.

DETAILED DESCRIPTION:
For the GWAS stage of this study, a cohort study will be conducted comparing hepatitis B patients with a response (see definitions below) versus patients who did not achieve a response to (peg)interferon treatment. Replication of SNPs identified by the GWAS will be performed in an independent cohort of patients with similar characteristics, treated with (peg)interferon. A large independent cohort of peginterferon treated HBV patients has already been identified guaranteeing a replication cohort.

ELIGIBILITY:
Inclusion criteria

* History of chronic hepatitis B, defined as the presence of positive hepatitis B surface antigen (HBsAg) for at least 6 months.
* History of treatment (per protocol or outside studies) with standard interferon (alfa-2a or alfa-2b), peginterferon alfa-2a or peginterferon alfa-2b for at least 12 weeks.
* A follow-up duration of at least 24 weeks after the last dose of (peg)interferon.
* Use of nucleos(t)ide analogues prior to or combined with (peg)interferon treatment is allowed.
* Available HBV DNA and HBeAg status at baseline, end of treatment and end of follow-up (24 weeks after end of treatment)
* Written informed consent obtained.

Exclusion criteria

* Co-infection with hepatitis C virus, delta virus or human immunodeficiency virus.
* Use of immunosuppressants, chemotherapy or systemic corticosteroids (prednisolone 30 mg daily or equivalent for more than 7 days) during (peg)interferon treatment or the 24-week pre- and post-treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients treated with (peg-)interferon
Sampling Method: Probability Sample
Enrollment: 1350 (Actual)
Dates: Start 2010-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Response to (PEG)IFN in relation to single-nucleotide polymorphisms identified by a GWAS | 24 weeks off-treatment
  Response:
  HBeAg-positive patients: HBV DNA <2000IU/ml and HBeAg seroconversion; 24 weeks off-treatment.
  HBeAg-negative patients: HBV DNA <2000IU/ml

SECONDARY OUTCOMES:
Response | 24 weeks off-treatment
  HBV DNA <20IU/ml for both HBeAg positives as negatives sustainability of HBeAg seroconversion or HBeAg loss(only HBeAg+ patients) HBsAg loss and seroconversion, ALT normalization, data on survival, incidence of cirrhosis, hepatocellular carcinoma and liver transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Harry LA Janssen, MD PhD, Principal Investigator — Foundation of Liver research (SLO), Rotterdam AND UHN liver clininc, Toronto Western & General Hospital; Pietro Lampertico, MD PhD, Study Chair — IRCCS Ca' Granda, Ospedale Maggiore Policlinico, University of Milan; Henry Chan, MD, Study Chair — The Chinese University of Hong Kong, Department of Medicine and Therapeutics; Jin-Lin Hou, MD PhD, Study Chair — Nanfang Hospital, Southern Medical University, Hepatology Unit and Dept of Infectious Diseases
Locations (1):
- Erasmus Medical Centre, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Brouwer WP, Chan HLY, Lampertico P, Hou J, Tangkijvanich P, Reesink HW, Zhang W, Mangia A, Tanwandee T, Montalto G, Simon K, Ormeci N, Chen L, Tabak F, Gunsar F, Flisiak R, Ferenci P, Akdogan M, Akyuz F, Hirankarn N, Jansen L, Wong VW, Soffredini R, Liang X, Chen S, Groothuismink ZMA, Santoro R, Jaroszewicz J, Ozaras R, Kozbial K, Brahmania M, Xie Q, Chotiyaputta W, Xun Q, Pazgan-Simon M, Oztas E, Verhey E, Montanari NR, Sun J, Hansen BE, Boonstra A, Janssen HLA; GIANT-B Global Consortium. Genome-wide Association Study Identifies Genetic Variants Associated With Early and Sustained Response to (Pegylated) Interferon in Chronic Hepatitis B Patients: The GIANT-B Study. Clin Infect Dis. 2019 Nov 13;69(11):1969-1979. doi: 10.1093/cid/ciz084. PMID 30715261